CLINICAL TRIAL: NCT00776516
Title: A Phase 1, Open-Label, Drug Interaction Study to Evaluate the Effect of Repeat Doses of Rifampin on the Single-Dose Pharmacokinetics of Mirabegron (YM178)
Brief Title: Pharmacokinetic Interaction Study to Assess the Effect of Repeat Doses of Rifampin on Mirabegron (YM178) in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: 178-CL-070
Record Dates: First submitted 2008-10-20; First posted 2008-10-21 (Estimated); Last update posted 2013-07-03 (Estimated); Status verified 2013-07

CONDITIONS: Pharmacokinetics of YM178
Keywords: Healthy volunteer subjects; CYP3A4 inducer; rifampin; drug interaction; pharmacokinetics; YM178; mirabegron
MeSH Terms: interventions — mirabegron; Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): mirabegron alone
  Interventions: Drug: mirabegron
- 2 (Experimental): mirabegron and rifampin
  Interventions: Drug: mirabegron; Drug: rifampin

INTERVENTIONS:
Drug: mirabegron — oral
  Other Names: YM178
Drug: rifampin — oral
  Other Names: Rifadin
  Arms: 2

SUMMARY:
The objective of the study is to assess the PK, safety and tolerability of a single dose of mirabegron alone and in combination with repeat doses of rifampin, a potent CYP3A4 inducer.

DETAILED DESCRIPTION:
A single group of patients will receive both mirabegron alone and in combination with rifampin

ELIGIBILITY:
Inclusion Criteria:

* Weighs at least 45 kg and body mass index (BMI) between 18 and 32 kg/m2 at Screening
* Normal or not clinically significant 12 lead ECG and clinical laboratory test results at Screening
* Female subjects must be post-menopausal, surgically sterile since at least 1 month prior to screening, or practicing effective non-hormonal contraceptive methods. All females must be non-lactating, and should have a negative result for the pregnancy test at Screening and on Day -1
* Negative drug and alcohol screens

Exclusion Criteria:

* Has known or suspected hypersensitivity to mirabegron or rifampin
* Liver enzyme test abnormalities (ALT, AST, or bilirubin) above the upper limit of normal
* History or presence of psychiatric illness, serious active or recurrent infection or hepatitis
* Previous history of cancer other than basal cell carcinoma or Stage 1 squamous cell carcinoma that has not been in remission for at least 5 years prior to the dose of study drug
* Donation or loss of ≥ 450 mL blood within 56 days prior to study drug administration or has donated plasma within 7 days prior to study drug administration
* Received or is anticipated to receive a prescription drug within 14 days prior to Day -1 or within 30 days prior to Day -1 for any long acting treatments. Use of any over-the-counter medications, including complementary and alternative medicines (except for occasional use of acetaminophen of up to 2000 mg/day but not more than 4 days per week) within 14 days prior to Day -1
* History of substance abuse within 6 months prior to Screening
* Current participation in another clinical trial or is taking or has been taking an investigational drug in the 30 days or 10 half lives of the drug, whichever is longer, prior to dosing
* Known to have hepatitis or HIV-1 and/or HIV-2 or is positive for hepatitis A antibody IgM, hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody at Screening
* Subject has consumed alcohol, caffeine-containing food or beverages, grapefruit juice, grapefruit-containing products or Seville oranges within 48 prior to Day -1

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2008-10; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Assess pharmacokinetics of mirabegron alone and in combination with rifampin | One month

SECONDARY OUTCOMES:
Assess safety and tolerability of mirabegron alone and in combination with rifampin | one month

CONTACTS AND LOCATIONS:
Overall Officials: Central Contact, Study Director — Astellas Pharma Global Development
Locations (1):
- Miami, Florida, United States

REFERENCES:
- [Background] Lee J, Moy S, Meijer J, Krauwinkel W, Sawamoto T, Kerbusch V, Kowalski D, Roy M, Marion A, Takusagawa S, van Gelderen M, Keirns J. Role of cytochrome p450 isoenzymes 3A and 2D6 in the in vivo metabolism of mirabegron, a beta3-adrenoceptor agonist. Clin Drug Investig. 2013 Jun;33(6):429-40. doi: 10.1007/s40261-013-0084-y. PMID 23625188